CLINICAL TRIAL: NCT05804513
Title: The Effect of Lixisenatide on the Effect of Pituitary Hormones
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tartu (Other)
Collaborators: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Vallo Volke, professor, University of Tartu
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Lixi22
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Healthy; Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sodium Chloride; Solutions; lixisenatide

STUDY DESIGN:
Intervention Model Description: Blinded randomised two group crossover
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo, healthy volunteers (Placebo Comparator): Sodium chloride 0.9% solution. Subcutaneous injection administered once.
  Interventions: Drug: Placebo
- Lixisenatide 10 micrograms, healthy volunteers (Active Comparator): Lixisenatide 10 micrograms. Subcutaneous injection administered once.
  Interventions: Drug: Lixisenatide 10 micrograms (50 micrograms/ml in 3 ml) Pen Injector
- Placebo, type 1 diabetic patients (Placebo Comparator): Sodium chloride 0.9% solution. Subcutaneous injection administered once.
  Interventions: Drug: Placebo
- Lixisenatide 10 micrograms, type 1 diabetic patients (Active Comparator): Lixisenatide 10 micrograms. Subcutaneous injection administered once.
  Interventions: Drug: Lixisenatide 10 micrograms (50 micrograms/ml in 3 ml) Pen Injector

INTERVENTIONS:
Drug: Placebo — s/c injection
  Other Names: Sodium chloride 0.9% solution
  Arms: Placebo, healthy volunteers; Placebo, type 1 diabetic patients
Drug: Lixisenatide 10 micrograms (50 micrograms/ml in 3 ml) Pen Injector — s/c injection
  Other Names: Lyxumia
  Arms: Lixisenatide 10 micrograms, healthy volunteers; Lixisenatide 10 micrograms, type 1 diabetic patients

SUMMARY:
The current study has two aims:

1. to test the hypothesis that a single dose of lixisenatide can be used as a growth hormone stimulation test;
2. to test if the growth hormone-stimulating effect is mediated by changes in blood glucose.

The secondary objective of the study is to monitor the effect of lixisenatide on other pituitary hormones and physiological parameters (blood glucose, blood pressure, heart rate, nausea).

DETAILED DESCRIPTION:
The randomized, blinded, placebo-controlled clinical trial is conducted on 5 healthy volunteers and 5 patients with type 1 diabetes.

All study subjects receive once a placebo and once 10 micrograms of lixisenatide.

The order of administration of study medication is decided on randomization. The placebo and lixisenatide are administered at least 2 days apart.

Blood samples are taken 30 minutes and immediately before study medication administration and 30, 60, 90, 120, and 150 minutes after study medication administration,.

The primary endpoint is the peak value of growth hormone measured during the 2,5 hours after study medication administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers:

   * male sex
   * age 18-60 years
   * body weight > 65 kg
2. Patients with type 1 diabetes:

   * type 1 diabetes
   * male sex
   * age 18-60 years
   * body weight > 65 kg
   * c-peptide in fasting blood sample <0,1 nmol/l
   * HbA1c < 8,5%

Exclusion Criteria:

1. Healthy volunteers:

   * use of aldosterone antagonist
   * use of glucocorticosteroid
   * use of other medication that potentially significantly affects pituitary function.
2. Patients with type 1 diabetes:

   * use of aldosterone antagonist
   * use of glucocorticosteroid
   * use of other medication that potentially significantly affects pituitary function.
   * The patient is excluded from the study if a significant change in blood glucose occurs in the study center.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Growth hormone area under the curve. | 0-150 minutes after study drug administration
  Treatment effect (placebo vs lixisenatide) on growth hormone area under curve (AUC) is compared between patients with type 1 diabetes and healthy volunteers.

SECONDARY OUTCOMES:
Growth hormone peak | 30, 60, 90, 120, and 150 minutes after the study drug administration.
  Maximum growth hormone concentration measured after study drug administration.
Glucose nadir | 30, 60, 90, 120, and 150 minutes after the study drug administration
  Lowest glucose concentration measured after the study drug administration
C-peptide peak | 30, 60, 90, 120, and 150 minutes after the study drug administration
  Maximum c-peptide concentration measured after the study drug administration
Cortisol peak | 30, 60, 90, 120, and 150 minutes after the study drug administration
  Maximum cortisol concentration measured after the study drug administration
Adrenocorticotropic hormone (ACTH) peak | 30, 60, 90, 120, and 150 minutes after the study drug administration
  Maximum ACTH concentration measured after the study drug administration
Prolactin peak | 30, 60, 90, 120, and 150 minutes after the study drug administration
  Maximum prolactin concentration measured after the study drug administration
Copeptin peak | 30, 60, 90, 120, and 150 minutes after the study drug administration
  Maximum copeptin concentration measured after the study drug administration
Aldosterone peak | 30, 60, 90, 120, and 150 minutes after the study drug administration
  Maximum aldosterone concentration measured after the study drug administration

OTHER OUTCOMES:
Nausea | 30, 60, 90, 120, and 150 minutes after the study drug administration
  The intensity of nausea on a 0-10 points visual analog scale, where 0 indicates no nausea and 10 worst imaginable nausea.
Systolic and diastolic blood pressure | 30, 60, 90, 120, and 150 minutes after the study drug administration
  The change in systolic and diastolic blood pressure compared to baseline.
Heart rate | 30, 60, 90, 120, and 150 minutes after the study drug administration.
  The change in heart rate compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Vallo Volke, MD, PhD, Principal Investigator — University of Tartu, Tartu University Hosptial
Locations (1):
- Tartu University Hospital, Tartu, Estonia